CLINICAL TRIAL: NCT00843791
Title: Ghrelin Regulation and Structure: Effect of Thiazolidinedione Therapy on Ghrelin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds to continue.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jonathan Purnell, Prinicipal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: eIRB 3941; OCTRI #10647 (Other: OCTRI); R01DK071161 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Insulin Resistance
Keywords: obesity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Treatment with placebo for 3 months before spectroscopy, hyperinsulinemic-euglycemic clamp, control diet, blood sampling.
  Interventions: Drug: placebo
- pioglitizone (Active Comparator): Treatment with pioglitazone for 3 months before hyperinsulinemic-euglycemic clamp, control diet with blood sampling and spectroscopy.
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: placebo — treatment with placebo for 3 months
  Arms: Placebo
Drug: pioglitazone — treatment with 30mg daily for two weeks then 45mg every day with pioglitazone for three months
  Other Names: thiazolidinedione therapy
  Arms: pioglitizone

SUMMARY:
The purpose of this study is to learn more about how insulin resistance (inability to process glucose correctly resulting in mildly elevated glucose levels) affects the hormone ghrelin.

DETAILED DESCRIPTION:
Insulin resistance suppresses fasting ghrelin levels and impairs postprandial ghrelin suppression. Improved insulin sensitivity with a thiazolidinedione will raise ghrelin levels, enhance meal-related suppression, but not change the ratio of total to active ghrelin or result in an alteration of ghrelin structure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80, weight stable for at least 3 months
* At lifetime maximal body weight and impaired glucose tolerance (ICT) by the World Health ORganization criteria:

  * fasting plasma glucose level of 100- 125mg/dL or
  * plasma glucose level between 140 to 149mg/dL following a 75gram oral glucose load

Exclusion Criteria:

* Actively losing weight
* Smokers
* Alcohol consumption > 2 drinks/day
* Prescription drug use
* Recreational drug use
* Type 2 Diabetes
* Conditions that contraindicate treatment with pioglitazone such as CHF, impaired liver or kidney function or known sensitivity to pioglitazone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited to participate in this aim from the Portland-Vancouver area through postings on the OHSU website, recruitment from previous studies, and advertisements in local newspapers. Original study recruitment dates were 2009 to 2013.
Pre-assignment Details: Following consent, patients undergo screening for entry criteria using blood work and an oral glucose tolerance test. Participants are excluded if they did not have impaired glucose tolerance and/or a contraindication to using a thiazolidinedione (pioglitazone or Actos), such as heart failure or abnormal liver studies.
Groups:
- Pioglitizone: Treatment with pioglitazone 30mg daily for two weeks then 45mg every day for 3 months before hyperinsulinemic-euglycemic clamp, control diet with blood sampling and spectroscopy.
Period: Overall Study
Arm/Group | Placebo | Pioglitizone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated early due to lack of funds.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitizone | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (5) | 40 (5.5) | 37 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Total and Active Ghrelin Levels
Description: The primary outcome of this study will be the comparison of ghrelin suppressibility (total and acylated) in response to meals obese subjects before and after 3-months therapy with a thiazolidinedione.
Time Frame: 0 and 3 months
Population: This aim was terminated early due to a shortage of funds and no samples were analyzed. There is no data to report
Groups:
- Pioglitizone: Treatment with pioglitizone (30 mg/45 mg) for 3 months before spectroscopy, hyperinsulinemic-euglycemic clamp, control diet, blood sampling.
Arm/Group | Placebo | Pioglitizone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 3 months per participant.
Groups:
- Pioglitazone: Treatment with pioglitazone for 3 months before spectroscopy, hyperinsulinemic-euglycemic clamp, control diet, blood sampling.
Arm/Group | Placebo | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Early termination due to fund shortage that led to small numbers of subjects enrolled and no measurements of primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No